CLINICAL TRIAL: NCT01426841
Title: Pilot Project of Adaptive Thoracic Radiotherapy for Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI Yee 25708
Record Dates: First submitted 2011-04-15; First posted 2011-09-01 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Small Cell Lung Cancer
Keywords: Small cell lung cancer; Adaptive radiotherapy; Thoracic radiotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Adaptive Radiation — Thoracic Radiotherapy which is adapted or adjusted during its course to account for tumor volume shrinkage which occurs during treatment

SUMMARY:
This study is intended to assess the feasibility of adjusting a radiation plan during its course to accommodate for a shrinking tumor target. The investigators hypothesize that an adaptive radiotherapy (RT) planning strategy for small cell lung cancer (SCLC) patients with chest-confined disease will allow for safe delivery of higher doses of chest RT than a non-adaptive RT planning approach without subjecting normal critical structures to unacceptable doses of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically or cytologically proven newly diagnosed small cell lung cancer
* chest-confined disease (including bulky intrathoracic disease)
* adequate pulmonary function tests (FEV-1>1.0 L, DLCO>50%)
* patients of childbearing potential must practice adequate contraception
* Age > or = 18 years
* Karnofsky performance status > or = 70
* eligible for concurrent chemoradiotherapy

Exclusion Criteria:

* patients who have undergone complete or subtotal tumour resection
* evidence of non-small cell histology
* prior or concurrent malignancy except non-melanomatous skin cancer unless disease-free for at least 5 years
* prior RT to the thorax or neck
* compromised lung function with inadequate pulmonary function tests (FEV-1<1.0,DLCO<50%)
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Differences in normal structure/target volume doses achievable using adaptive radiotherapy approach | 12-24 months
  Differences in normal structure/target volume doses achievable using adaptive radiotherapy approach will be measured in centigray

SECONDARY OUTCOMES:
Local control and patterns of failure | 12-24 months
  Local control and patterns of failure
Survival | 12-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Don Yee, MD, FRCPC, Principal Investigator — Cross Cancer Institute, Alberta Health Services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada